CLINICAL TRIAL: NCT04323410
Title: Casting in Finger-trap Traction Without Reduction Versus Closed Reduction and Percutaneous Pin Fixation of Dorsally Displaced, Overriding Distal Metaphyseal Radius Fractures in Under Eleven Years Old Children
Brief Title: Casting Versus Percutaneus Pinning Treatment of Pediatric Overriding Distal Forearm Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Topi Laaksonen, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PediatricOverridingFractures
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Pediatric Overriding Distal Metaphyseal Radius Fractures
Keywords: bayonet fracture; paediatric fracture; distal forearm fracture; overriding fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast immobilization (Experimental): In the casting group, padded synthetic dorsal above elbow and volar below elbow splints are applied in ED without local or general anesthesia. Dorsal displacement and shortening of the radius are not corrected, but the forearm is attempted to be manipulated straight during application of the splints. The casted forearm is then supported by a collar and cuff sling. Splints are removed in an outpatient clinic at 4 weeks.
  Cast immobilization is discontinued after 4 weeks and when the fracture site is nontender. If palpated tenderness is still present, the patient is given a dorsal forearm splint which can be removed (maximum of 2 weeks usage).
  Interventions: Procedure: Cast immobilization
- Percutaneus pinning (Active Comparator): In the surgery group, a padded dorsal above elbow splint is applied in ED. Reduction and percutaneous pinning are performed under anesthesia in operating room by an experienced attending pediatric orthopedic surgeon within 7 days from the injury. Pin fixation is performed with two 1.6 mm pins. Padded dorsal above elbow and volar below elbow splints are applied. Splints and pins are removed at the outpatient clinic at 4 weeks after surgery.
  Interventions: Procedure: Percutaneus pinning

INTERVENTIONS:
Procedure: Cast immobilization — Cast immobilisation is done using finger trap traction. The fractured forearm is splinted above elbow with dorsal cast without attempted reduction.
  Arms: Cast immobilization
Procedure: Percutaneus pinning — Reduction under fluoroscopic guidance and fixation using two crossing 1.6mm K-wires.
  Arms: Percutaneus pinning

SUMMARY:
This is a randomized controlled trial comparing casting in finger-trap traction without reduction versus closed reduction and percutaneous pin fixation of dorsally displaced, overriding distal metaphyseal radius fractures in under eleven years old children.

DETAILED DESCRIPTION:
Overriding pediatric distal radius fractures have been managed with anatomical reduction performed under anesthesia with or without percutaneous pinning. This research protocol was developed due to good results reported on leaving the fractures in an overriding position.

In this randomized controlled trial, we will compare objective outcomes between casting in finger-trap traction without reduction versus closed reduction and percutaneous pin fixation of dorsally displaced, overriding distal metaphyseal radius fractures in children.

Inclusion criteria are patients younger than 11 years old (Tanner 0) with completely overriding distal radius fractures. At the emergency department patients are randomized into two groups: finger trap traction and cast immobilization (experimental group) and anatomic reduction and percutaneous pin fixation (control group).

The current controversy is whether cast immobilization alone is an adequate stabilization or whether percutaneous pin fixation is more appropriate for displaced, complete, distal forearm (overriding) metaphyseal fractures. The objectives of this trial are to compare the outcomes between conservative treatment with finger trap method for completely displaced distal radius fractures and surgical treatment with percutaneous pinning. Our null hypothesis is that there are no radiological or clinically relevant differences in outcome measures between the two treatment groups. We consider non-inferiority proven if there is no clinically significant difference at 6 months between the two treatments groups in the primary outcome: ratio (%) of forearm rotation and wrist extension-flexion range of motion (ROM) compared to the non-affected side at 6 months (non-inferiority margin 10%).

ELIGIBILITY:
Inclusion Criteria:

* Child with open epiphysis with closed overriding metaphyseal distal radial fracture with or without an associated fracture of the ulna
* Normal communication development (languages Finnish, Swedish, English)

Exclusion Criteria:

* Bilateral forearm injuries
* Gustillo-Anderson grade II or III open fracture
* Galeazzi fracture-dislocation
* Polytrauma
* Neurovascular injury of the ipsilateral upper extremity
* History of a displaced forearm fracture
* Underlying disease affecting fracture healing

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wrist ROM | 6 months
  The ratio (injured side/non-injured side) in total active range of motion of the wrist in the flexion-extension plane.
Forearm ROM | 6 months
  The ratio (injured side/non-injured side) in the total active forearm rotation.

SECONDARY OUTCOMES:
Patient-reported pain | 1 and 4 weeks, 3 and 6 months, 1 year
  Pain at rest and in activities is assessed on PedsQL questionnaire. Range 0 to 100 mm, 0 best.
Patient-reported outcome (PROM) | 4 weeks, 3 and 6 months, 1 year
  Quick-DASH, range 0 to 100, 0 best
Radiographic outcomes | 1 and 4 weeks, 3 and 6 months, 1 year
  Sagittal and coronal plain radiographs
Grip strength | 3 and 6 months, 1 year
  Objective grip strength measurement using dynamometer
Forearms length | 3 and 6 months, 1 year
  Length of forearms and hands
Wrist ROM | 3 months, 1 year
  The ratio (injured side/non-injured side) in total active range of motion of the wrist in the flexion-extension plane.
Forearm ROM | 3 months, 1 year
  The ratio (injured side/non-injured side) in the total active forearm rotation.
Overall satisfaction | 6 months
  The patient's parent(s) or guardian(s) are queried about their satisfaction with the treatment. The satisfaction of the function of the fractured upper extremity and its effect on the patient's daily living and satisfaction to the cosmetic outcome are recorded on a 5-step Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- New Children's Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laaksonen T, Stenroos A, Puhakka J, Kosola J, Kautiainen H, Ramo L, Nietosvaara Y. Casting in finger trap traction without reduction versus closed reduction and percutaneous pin fixation of dorsally displaced, over-riding distal metaphyseal radius fractures in children under 11 years old: a study protocol of a randomised controlled trial. BMJ Open. 2021 May 26;11(5):e045689. doi: 10.1136/bmjopen-2020-045689. PMID 34039573